CLINICAL TRIAL: NCT00779714
Title: Prospectively Randomized Phase III Study of an Individualized Sensitivity-Directed Combination Chemotherapy Versus DTIC as First-Line Treatment in Stage IV Metastatic Melanoma
Brief Title: Comparative Study of Individualized Sensitivity-Directed Chemotherapy Versus DTIC
Acronym: ChemoSensMM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Collaborators: Hiege-Stiftung gegen Hautkrebs (Unknown); medac GmbH (Industry); DCS Innovative Diagnostik Systeme (Unknown)
Responsible Party: Prof. Dr. med. Selma Ugurel, Dept of Dermatology, University of Wuerzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101.321-13/07; EudraCT Nr. 2008-001686-28
Record Dates: First submitted 2008-10-22; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Melanoma
Keywords: metastatic (AJCC stage IV); first-line chemotherapy; ex-vivo chemosensitivity profiling; evaluation of biomarkers
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Dacarbazine; TP protocol; treosulfan; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (individualized combined chemotherapy) (Experimental)
  Interventions: Drug: paclitaxel + cisplatin; Drug: treosulfan + cytarabine
- B (DTIC monochemotherapy) (Active Comparator)
  Interventions: Drug: DTIC (dacarbazine)

INTERVENTIONS:
Drug: DTIC (dacarbazine) — 1000 mg/m2, d1 every 21 days
  Other Names: detimedac
  Arms: B (DTIC monochemotherapy)
Drug: paclitaxel + cisplatin — paclitaxel 200 mg/m2 cisplatin 50 mg/m2 d1 every 21 days
  Other Names: taxomedac + cisplatin medac
  Arms: A (individualized combined chemotherapy)
Drug: treosulfan + cytarabine — treosulfan 2500 mg/m2, d2 cytarabine 100 mg/m2, d1-3 every 21 days
  Other Names: ovastat + alexan
  Arms: A (individualized combined chemotherapy)

SUMMARY:
This phase III trial is aimed to investigate the efficacy of an individualized, sensitivity-directed combination chemotherapy in comparison to the standard regimen DTIC.

Two question are aimed to be answered by this study:

1. Is the individual chemosensitivity index (BICSI) a prognostic / predictive biomarker for chemotherapy ?
2. Is an individualized, sensitivity-directed combination chemotherapy superior to the standard regimen DTIC in terms of survival and response ?

DETAILED DESCRIPTION:
Melanoma is a cutaneous neoplasm known for its high aggressiveness, its early dissemination of metastases, and its poor prognosis once metastasized. Chemotherapy with dacarbacine (DTIC) is widely accepted as the standard treatment in metastatic melanoma, with reported response rates of about 10%. This poor outcome is assumed to be due to a high chemoresistance intrinsic to melanoma cells. However, other therapeutic options like polychemotherapy, biochemotherapy, immunotherapy as well as targeted agents did not yet prove to be superior to DTIC in multicenter randomized studies.

Therefore, chemotherapy still is considered as the main therapeutic option in advanced metastatic melanoma, and a number of non-standard chemotherapeutics have been tested in small pilot studies to improve treatment efficacy. Even though complete remissions of metastatic lesions could only be observed in a few patients, these observations indicate a subgroup of patients exhibiting high sensitivity to certain anticancer drugs. An in vitro ATP-based chemosensitivity assay has been shown to differentiate between chemosensitive and chemoresistant melanoma patients. A phase-II-study testing this assay in 53 metastatic melanoma patients followed by a sensitivity-directed individualized chemotherapy demonstrated, that the chemosensitivity profile of an individual patient, reflected by the best individual chemosensitivity index (BICSI), correlated with therapy outcome in terms of therapy response and patient overall survival (Ugurel S: Clin Cancer Res 2006). Interestingly, a surprisingly high proportion of about 2/5 of the investigated patient cohort were classified as chemosensitive, the remaining 3/5 were classified as chemoresistant. Objective response was 36.4% in chemosensitive patients compared to 16.1% in chemoresistant patients (p=0.114); progression arrest (CR+PR+SD) was 59.1% versus 22.6% (p=0.01). Chemosensitive patients showed an increased overall survival of 14.6 months compared to 7.4 months in chemoresistant patients (p=0.041).

These encouraging results prompted the initiation of this randomized phase-III-trial investigating an individualized sensitivity-directed combination chemotherapy compared to the current standard treatment DTIC, as first-line treatment in metastatic melanoma. The therapeutics for chemosensitivity testing and treatment of patients were chosen considering the results of the phase-II-trial (paclitaxel+cisplatinum, treosulfan+cytarabine).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma of the skin, mucosa, or unknown primary, diagnosed with surgically unresectable distant metastases (stage IV according to AJCC).
* At least one measurable target lesion according to RECIST, assessed by CT or MRI (tumor assessment by X-ray or ultrasonography only is not allowed).
* Access to a biopsy of ~1 cm3 from at least one metastatic lesion for in vitro chemosensitivity testing. Cell suspensions from malignant effusions are also eligible.
* No prior chemotherapy in stage IV (adjuvant chemotherapy in stage III allowed; one prior regimen of immunotherapy or targeted therapy in stage IV allowed).
* No evidence of brain/CNS metastases. Former history of brain/CNS metastases, which have been treated successfully, and are no longer visible in CT/MRI is allowed.
* Last complete tumor assessment (CT or MRI of thorax, abdomen and brain) not older than 14 days prior to registration, and not older than 5 weeks prior to onset of study treatment.
* ECOG/WHO performance index of 0 or 1.
* Patients must have stopped any kind of previous antineoplastic therapy for at least 2 weeks prior to registration, and at least 4 weeks prior to treatment onset.
* Patients must not have concurrent or recent malignancies except for surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin. Patients with previous malignancies, which have been treated with a subsequent disease-free interval of at least 5 years, are eligible.
* Patient age ≥ 18 years.
* Adequate hematological, renal and liver function as defined by the following laboratory values performed within 14 days prior to randomisation:

  * absolute neutrophil count (ANC) ≥ 1.5 x 109/l
  * platelet count ≥ 100 x 109/l
  * hemoglobin ≥ 9 g/dl
  * urea and serum creatinine ≤ 2 times upper normal limit (UNL)
  * total and direct serum bilirubin ≤ 2 times UNL
  * GOT or GPT ≤ 2.5 times UNL; ≤ 5 times UNL is allowed in case of liver metastasis
  * alkaline phosphatase < 2.5 times UNL
* Female patients should not be pregnant or nursing. Women of childbearing potential should be using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner). For subjects using a hormonal contraceptive method, information regarding the product under evaluation and its potential effect on the contraceptive should be addressed.
* Male patients should use an effective method of contraception.
* Before registration, written informed consent must be given according to GCP guidelines and national/local regulations. Patients must be willing and giving informed consent to participation in the trial.

Exclusion Criteria:

* All metastatic lesions are surgically resectable.
* Prior chemotherapy in stage IV (adjuvant chemotherapy in stage III allowed; one prior regimen of immunotherapy or targeted therapy in stage IV allowed).
* Primary melanoma of the uvea / choroidea.
* Evidence of brain/CNS metastases. Former history of brain/CNS metastases, which have been treated successfully, and are no longer visible in CT/MRI is allowed.
* ECOG/WHO performance index of 2 or higher
* Concurrent or recent malignancies except for surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin. Patients with previous malignancies, which have been treated with a subsequent disease-free interval of at least 5 years, are eligible.
* Any severe or uncontrolled hematological, renal or liver dysfunction as defined by the laboratory values given in Inclusion Criteria.
* Any clinically uncontrolled infectious disease including HIV positivity or AIDS-related illness.
* Any female patients who are pregnant or nursing.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Disease-specific overall survival | 4 years

SECONDARY OUTCOMES:
Objective response | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Selma Ugurel, Prof. (MD), Study Chair — Dept of Dermatology, University of Wuerzburg
Locations (23):
- Germany (23):
  - Dept of Dermatology, University of Aachen, Aachen
  - Dept of Dermatology, University of Berlin Charite, Berlin
  - Dept of Dermatology, University of Bochum, Bochum
  - Medizinisches Zentrum Bonn Friedensplatz, Bonn
  - Dept of Dermatology, University of Essen, Essen
  - Dermatology, Klinikum Frankfurt/Oder, Frankfurt (Oder)
  - Dept of Dermatology, University of Frankfurt, Frankfurt am Main
  - Dept of Dermatology, University of Hannover, Hanover
  - Dept of Dermatology, Saarland University, Homburg/Saar
  - Dept of Dermatology, University of Jena, Jena
  - Dept of Dermatology, University of Schleswig-Holstein Campus Kiel, Kiel
  - Dermatology, Klinikum Ludwishafen, Ludwigshafen
  - Dept of Dermatology, University of Schleswig-Holstein Campus Luebeck, Lübeck
  - Dept of Dermatology, Univeristy of Magdeburg, Magdeburg
  - Dept of Dermatology, University of Mainz, Mainz
  - Dept of Dermatology, University of Mannheim, Mannheim
  - Dept of Dermatology, University of Marburg, Marburg
  - Dept of Dermatology, University of Muenchen, München
  - Dept of Dermatology, University of Muenster, Münster
  - Dept of Medical Oncology, Fachklinik Hornheide, Münster
  - Dermatology, Klinikum Dorothea Christiane Erxleben, Quedlinburg
  - Dept of Dermatology, University of Tuebingen, Tübingen
  - Dept of Dermatology, University of Wuerzburg, Würzburg

REFERENCES:
- [Background] Ugurel S, Schadendorf D, Pfohler C, Neuber K, Thoelke A, Ulrich J, Hauschild A, Spieth K, Kaatz M, Rittgen W, Delorme S, Tilgen W, Reinhold U; Dermatologic Cooperative Oncology Group. In vitro drug sensitivity predicts response and survival after individualized sensitivity-directed chemotherapy in metastatic melanoma: a multicenter phase II trial of the Dermatologic Cooperative Oncology Group. Clin Cancer Res. 2006 Sep 15;12(18):5454-63. doi: 10.1158/1078-0432.CCR-05-2763. PMID 17000680
- [Background] Ugurel S, Tilgen W, Reinhold U. Chemosensitivity testing in malignant melanoma. Recent Results Cancer Res. 2003;161:81-92. doi: 10.1007/978-3-642-19022-3_8. PMID 12528801
- [Background] Cree IA, Neale MH, Myatt NE, de Takats PG, Hall P, Grant J, Kurbacher CM, Reinhold U, Neuber K, MacKie RM, Chana J, Weaver PC, Khoury GG, Sartori C, Andreotti PE. Heterogeneity of chemosensitivity of metastatic cutaneous melanoma. Anticancer Drugs. 1999 Jun;10(5):437-44. doi: 10.1097/00001813-199906000-00002. PMID 10477162
- [Background] Andreotti PE, Cree IA, Kurbacher CM, Hartmann DM, Linder D, Harel G, Gleiberman I, Caruso PA, Ricks SH, Untch M, et al. Chemosensitivity testing of human tumors using a microplate adenosine triphosphate luminescence assay: clinical correlation for cisplatin resistance of ovarian carcinoma. Cancer Res. 1995 Nov 15;55(22):5276-82. PMID 7585588
- See also: Homepage of organization (ADO, DeCOG) conducting this trial — http://www.ado-homepage.de